CLINICAL TRIAL: NCT04392492
Title: Plug-based Percutaneous Vascular Closure Device in Transcatheter Aortic Valve Replacement
Brief Title: Vascular Closure Device in Transcatheter Aortic Valve Replacement
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Dalén, Associate professor, Karolinska University Hospital
Other Study IDs: MANTA TAVI
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients undergoing transfemoral TAVI with MANTA closure: Patients undergoing transfemoral transcatheter aortic valve replacement with femoral access site closure using the novel plug-based vascular closure device (MANTA, Teleflex/Essential Medical Inc., Malvern, Pennsylvania, USA).
  Interventions: Device: MANTA vascular closure device

INTERVENTIONS:
Device: MANTA vascular closure device — Femoral access site closure using the MANTA closure device

SUMMARY:
Evaluation of the safety and efficacy of a percutaneous plug-based large-bore vascular closure device for femoral artery closure in an unselected consecutive patient cohort undergoing transcatheter aortic valve implantation in a single-center prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing transfemoral TAVI at the Karolinska University Hospital

Exclusion Criteria:

* Patients undergoing TAVI with access other than transfemoral
* Use of closure device other than MANTA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients undergoing TAVI at the Karolinska University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-25 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with major vascular complications | 6 week follow up
  Major vascular access site complications according to the VARC-2 definitions

SECONDARY OUTCOMES:
Number of patients with minor vascular complications | 6 week follow up
  Minor vascular access site complications according to the VARC-2 definitions
Number of patients with vascular closure device failure | 6 week follow up
  Percutaneous vascular closure device failure according to the VARC-2 definitions
Number of patients with life-threatening, disabling or major bleeding | 6 week follow up
  Life-threatening, disabling or major bleeding complications according to the BARC definitions

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Kastengren M, Settergren M, Ruck A, Feldt K, Saleh N, Linder R, Verouhis D, Meduri CU, Bager J, Dalen M. Percutaneous plug-based vascular closure device in 1000 consecutive transfemoral transcatheter aortic valve implantations. Int J Cardiol. 2022 Jul 15;359:7-13. doi: 10.1016/j.ijcard.2022.04.033. Epub 2022 Apr 12. PMID 35427700